CLINICAL TRIAL: NCT07121803
Title: Analysis of Effects of Specialized Food Products Based on Ice-Cream on Esophageal Motility
Brief Title: The Influence of Specialized Food Products Based on Ice-Cream on Esophageal Motility
Acronym: MICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Russian Science Foundation (Other); Group of companies EFKO (Unknown)
Responsible Party: Principal Investigator, Sergey Morozov, Principal Investigator, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OGIG-2025-MICE
Record Dates: First submitted 2025-08-01; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Ineffective Esophageal Motility; GERD (Gastroesophageal Reflux Disease)
Keywords: Esophageal motility; Specialized foods; icecream; esophagus; motility; high-resolution esophageal manometry
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Ice Cream; maltitol; oligofructose; Inulin; Erythritol

STUDY DESIGN:
Intervention Model Description: This is a double-blind cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Subjects of this arm will receive the following sequence of products: 1 - ice cream with brazzein, maltitol and oligofructose, 2 - ice cream with brazzein, erythritol, maltitol and inulin; 3 - standard ice cream
  Interventions: Other: specialized food based on ice cream, order 1
- Arm 2 (Experimental): Subjects of this arm will receive the following sequence of products: 1 - ice cream with brazzein, erythritol, maltitol and inulin; 2 - ice cream with brazzein, maltitol and oligofructose, 3 - standard ice cream
  Interventions: Other: specialized food based on ice cream, order 2
- Arm 3 (Experimental): Subjects of this arm will receive the following sequence of products: 1 - standard ice cream; 2 - ice cream with brazzein, maltitol and oligofructose, 3 - ice cream with brazzein, erythritol, maltitol and inulin
  Interventions: Other: specialized food based on ice cream, order 3

INTERVENTIONS:
Other: specialized food based on ice cream, order 1 — Order of intervention: 1. ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose; 2: ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin; 3: standard ice cream (12% fat)
  Other Names: specialized food product based on ice cream; ice cream with brazzein, maltitol and oligofructose; ice cream with brazzein, maltitol, inulin, erythritol; standard ice cream (sundae)
  Arms: Arm 1
Other: specialized food based on ice cream, order 2 — 1. ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin;
  2. ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose;
  3. standard ice cream (12% fat)
  Arms: Arm 2
Other: specialized food based on ice cream, order 3 — 1. standard ice cream (12% fat)
  2. ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose
  3. ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin
  Arms: Arm 3

SUMMARY:
This study aims to assess the influence of specialized products based on ice cream on esophageal motility

DETAILED DESCRIPTION:
During this study participants will be examined with the use of high-resolution esophageal motility. After standard procedure, according to Chicago IV protocol, subjects will be provided with 3 different types of food products: standard icecream (sundae), icecream with brazzein, maltitol and oligofructose; icecream with brazzein, erythritol, maltitol and inulin. Tolerability of products will be assessed based on specialized scales and formal questioning.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate based on signed written informed consent;
* controlled glycemia. If stable glycemia is achieved on treatment, the following requirements should be met:
* no qualitative changes in treatment within 6 months before enrollment (i.e., the introduction of a new antidiabetic therapy);
* doses of anti-diabetic medications should be stable for 6 month in patients who receive metformin, gliptins, sulfonylureas, sodium/glucose cotransporter 2 (SGLT-2) inhibitors, glucagon-like peptide 1 agonists (GLP-1) or insulin.
* no new medications during participation in the study

Exclusion Criteria:

* Pregnancy and breastfeeding;
* Liver cirrhosis based on liver histology, or liver stiffness measurement (LSM > or = 14 kPa by Fibroscan), or APRI > or= 1; or BARD score > or = 2.
* Diarrhea of any type (watery stool more than 3 times a day).
* Chronic heart failure (I-IV class by NYHA).
* Past major abdominal or chest surgery, including bariatric procedures and fundoplication (except appendectomy or cholecystectomy performed more than a year before enrollment).
* Achalasia and esophago-gastric junction outflow obstruction
* Major esophageal motility disorders according to Chicago IV classification.
* Clinically relevant acute cardiovascular event within 6 months prior to screening.
* Uncontrolled arterial hypertension despite optimal anti-hypertensive therapy.
* Diabetes mellitus type 1.
* The level of glycated hemoglobin [HbA1c] >9.0%.
* Hypersensitivity to the studied product or any of its components, including lactose intolerance.
* The intake of any pharmaceutical agents with known influence on esophageal motility (including, but not limited to: beta-blockers, calcium channel blockers, m-cholinoblockers, myorelaxants, antidepressants, tranquilizers, prokinetic agents)
* Any medical conditions that may significantly affect life expectancy, including known cancers;
* Any clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, tumor or psychiatric diseases;
* Mental instability or incapacity, which may impact the ability to give informed consent, take part in the study, or affect the ability to comply with the requirements of the study protocol;
* Inability to tolerate high-resolution esophageal manometry without sedation, at least in part.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean lower esophageal sphincter resting pressure | baseline, during the intervention
  Based on the high-resolution esophageal manometry measurement
Distal contractile integral | baseline, during the intervention
mean lower esophageal sphincter integral relaxation pressure | baseline, during the intervention
  IRP 4
Mean contractile front velocity | baseline, during the intervention
  CFV
Distal latency | baseline, during the intervention
  DL
Mean intrabolus pressure | baseline, during the intervention
  IBP

SECONDARY OUTCOMES:
mean upper esophageal sphincter resting pressure | baseline, during the intervention
  mean UES resting pressure
Mean upper esophageal sphincter integrated relaxation pressure | baseline, during the intervention
  Mean UES IRP 2 sec
product organoleptic assessment | during the intervention
  organoleptic assessment on taste, scent, colour and texture with the use of a special form based on visual-analogue scale (range: 1 - 5, where 1 is worse assessment, and 5 - favourable assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Morozov, MD, PhD, Principal Investigator — Federal Research Center of Nutrition and Biotechnology
Locations (1):
- Dpt Gastroenterology, Hepatology and Nutrition, Federal Research Centre of Nutrition and Biotechnology, Kashirskoye shosse, bld 21, Moscow, Russia., Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared upon reasonable request to PI
Supporting Information: Study Protocol, ICF, CSR
Time Frame: within 2 years upon study completion
Access Criteria: Qualified persons who applied reasonable request to access the data. According to the local law, only depersonalized data may be shared.
URL: https://ion.ru